CLINICAL TRIAL: NCT01570543
Title: Development of MR Systems, Accessories, and Software for Imaging Subjects With Metallic Orthopedic Implants.
Brief Title: MRI Scanning of People With MR Safe Orthopedic Implants That Are Made of Metal
Acronym: MRI
Status: Withdrawn | Type: Observational
Why Stopped: After over a year no subjects were identified
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 114-2011-GES-0029
Record Dates: First submitted 2012-03-13; First posted 2012-04-04 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2012-10

CONDITIONS: Implants
Keywords: implants; knee implants; hip implants; metallic implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- orthopedic implants, no treatment

SUMMARY:
The purpose of the study is to improve image quality, increase speed of scanning and to see how well certain products test by scanning people who have an orthopedic hip or knee metallic implant.

DETAILED DESCRIPTION:
The technology comprising Magnetic Resonance (MR) imaging systems and accessories is under continuous development in order to improve the quality of images, speed of acquisition, and usability of MR devices applied to image subjects with metallic orthopedic implants. Collection of in vivo human data throughout the product development and maintenance lifecycle plays an important role in enabling the technology to be investigated, optimized, and validated.

This is a pre-market investigation involving commercially available devices, investigational devices, and commercial devices modified with investigational components. The Study will be conducted for three years, over which time a number of endpoints will be collected for various devices under development.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age; and
* Must have an in-place knee or hip orthopedic implant; and
* Must have a metallic orthopedic implant that is labeled as "MR safe" or "MR Conditional" by the implant manufacturer; and
* Must be able to provide sufficient documentation of the implant such that study staff can confirm its compatibility with the specific MR environment per the implant labeling; and
* Must be able to provide written documentation or attestation of the date their orthopedic implant was placed; and
* Must be able to hear and understand English without assistive devices; and
* Must provide written informed consent; and
* Must provide the name and contact information for his/her Physician

Exclusion Criteria:

* Any implant more than 5 years old
* Any implant that is investigational
* Any implant which cannot be verified with a manufacturer's label
* Any implant implanted outside of U.S.A.
* Any implant associated with a recall
* Any history of pathology associated with an in-place orthopedic implant
* History of pain at implant site, in the past 30 days
* Known or suspected complication, defect, or concern regarding an in-place orthopedic implant
* Surgery related to an orthopedic implant within the past 120 days
* Potential for metal to be in body due to a previous injury involving metallic objects
* Pregnancy or late menstrual period
* Any non-orthopedic implant
* Any type of prosthesis (eye, penile, heart valve, etc.)
* Any other type of metal implant other than knee or hip implant
* Presence of tissue expander (breast)
* Intra-uterine device, diaphragm or pessary
* Loose dental fillings or dental fillings in the last 30 days
* Tattoo or permanent make up
* Breathing problem or motion disorder
* Claustrophobia or panic attacks
* Hearing Aid
* Body piercing jewelry
* Dentures or partial plates
* External medical hardware (example: orthopedic braces, orthodontic appliance)
* Known or past allergic reactions to latex

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample from Waukesha, Wisconsin area.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Image quality of images that are obtained from scanning subjects who have metallic MR Safe or MR Conditional implants, will be evaluated on a pass/fail basis. | Within the first hour after scanning
  Review of real-time and post-acquisition technical assessment will occur. The assessment of images will be made by scientists, engineers and radiology technologists. Validation activities will consist of a comparison of the observed images with the prospective acceptance criteria to determine if each specific test results in a pass or fail. There are no statistical tests and no efficacy endpoints.

SECONDARY OUTCOMES:
The ease of use and optimization of the MR device in imaging of subjects with metallic implants will be assessed. | Within one hour of scanning
  Software programs, data processing software and other types of MR system accessory hardware and software components will be tested and evaluated for how easy and problem-free they are to use and optimize for imaging of subjects with a metallic implant. Once this is established, validation of user requirements and specifications will be performed in accordance with Good Manufacturing Practice (GMP) design control requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Lewein, Principal Investigator — American Registry of Radiologic Technologists
Locations (1):
- GE Healthcare, Waukesha, Wisconsin, United States

REFERENCES:
- [Background] Nyenhuis, J. A., Kildishev, A. V., Athey, T. W., Bourland, J. D., Foster, K. S., Graber, G. P., "Heating Near Implanted Medical Devices by the MRI RF-magnetic Field," IEEE Trans. Magn., Vol 35, 1999, pp. 4133-4135
- [Background] Potter HG, Nestor BJ, Sofka CM, Ho ST, Peters LE, Salvati EA. Magnetic resonance imaging after total hip arthroplasty: evaluation of periprosthetic soft tissue. J Bone Joint Surg Am. 2004 Sep;86(9):1947-54. doi: 10.2106/00004623-200409000-00013. PMID 15342757
- [Background] Hayter CL, Koff MF, Shah P, Koch KM, Miller TT, Potter HG. MRI after arthroplasty: comparison of MAVRIC and conventional fast spin-echo techniques. AJR Am J Roentgenol. 2011 Sep;197(3):W405-11. doi: 10.2214/AJR.11.6659. PMID 21862766
- [Background] Cook SM, Pellicci PM, Potter HG. Use of magnetic resonance imaging in the diagnosis of an occult fracture of the femoral component after total hip arthroplasty. A case report. J Bone Joint Surg Am. 2004 Jan;86(1):149-53. doi: 10.2106/00004623-200401000-00024. No abstract available. PMID 14711959
- [Background] Sofka CM, Potter HG. MR imaging of joint arthroplasty. Semin Musculoskelet Radiol. 2002 Mar;6(1):79-85. doi: 10.1055/s-2002-23166. PMID 11917273
- [Background] Suh JS, Jeong EK, Shin KH, Cho JH, Na JB, Kim DH, Han CD. Minimizing artifacts caused by metallic implants at MR imaging: experimental and clinical studies. AJR Am J Roentgenol. 1998 Nov;171(5):1207-13. doi: 10.2214/ajr.171.5.9798849.
- [Background] Henk CB, Brodner W, Grampp S, Breitenseher M, Thurnher M, Mostbeck GH, Imhof H. The postoperative spine. Top Magn Reson Imaging. 1999 Aug;10(4):247-64. doi: 10.1097/00002142-199908000-00006. PMID 10616816
- [Background] Hayter CL, Koff MF, Potter HG. Magnetic resonance imaging of the postoperative hip. J Magn Reson Imaging. 2012 May;35(5):1013-25. doi: 10.1002/jmri.23523. PMID 22499278
- [Background] Koch KM, Lorbiecki JE, Hinks RS, King KF. A multispectral three-dimensional acquisition technique for imaging near metal implants. Magn Reson Med. 2009 Feb;61(2):381-90. doi: 10.1002/mrm.21856. PMID 19165901
- [Background] Koch KM, Brau AC, Chen W, Gold GE, Hargreaves BA, Koff M, McKinnon GC, Potter HG, King KF. Imaging near metal with a MAVRIC-SEMAC hybrid. Magn Reson Med. 2011 Jan;65(1):71-82. doi: 10.1002/mrm.22523. PMID 20981709
- [Background] Koch KM, Hargreaves BA, Pauly KB, Chen W, Gold GE, King KF. Magnetic resonance imaging near metal implants. J Magn Reson Imaging. 2010 Oct;32(4):773-87. doi: 10.1002/jmri.22313. PMID 20882607
- [Background] Potter HG, Foo LF. Magnetic resonance imaging of joint arthroplasty. Orthop Clin North Am. 2006 Jul;37(3):361-73, vi-vii. doi: 10.1016/j.ocl.2006.03.003. PMID 16846767
- [Background] Walde TA, Weiland DE, Leung SB, Kitamura N, Sychterz CJ, Engh CA Jr, Claus AM, Potter HG, Engh CA Sr. Comparison of CT, MRI, and radiographs in assessing pelvic osteolysis: a cadaveric study. Clin Orthop Relat Res. 2005 Aug;(437):138-44. doi: 10.1097/01.blo.0000164028.14504.46. PMID 16056041
- [Background] Weiland DE, Walde TA, Leung SB, Sychterz CJ, Ho S, Engh CA, Potter HG. Magnetic resonance imaging in the evaluation of periprosthetic acetabular osteolysis: a cadaveric study. J Orthop Res. 2005 Jul;23(4):713-9. doi: 10.1016/j.orthres.2005.02.007. Epub 2005 Apr 12. PMID 16022981
- [Background] Hayter CL, Potter HG, Su EP. Imaging of metal-on-metal hip resurfacing. Orthop Clin North Am. 2011 Apr;42(2):195-205, viii. doi: 10.1016/j.ocl.2010.12.006. PMID 21435495
- [Background] Hayter CL, Potter HG, Padgett DE, Perino G, Nestor BJ. MRI assessment of wear-induced synovitis. ISMRM Annual Conference, paper presentation. Montreal; 2011.
- [Background] Campbell P, Ebramzadeh E, Nelson S, Takamura K, De Smet K, Amstutz HC. Histological features of pseudotumor-like tissues from metal-on-metal hips. Clin Orthop Relat Res. 2010 Sep;468(9):2321-7. doi: 10.1007/s11999-010-1372-y. PMID 20458645
- [Background] Pandit H, Glyn-Jones S, McLardy-Smith P, Gundle R, Whitwell D, Gibbons CL, Ostlere S, Athanasou N, Gill HS, Murray DW. Pseudotumours associated with metal-on-metal hip resurfacings. J Bone Joint Surg Br. 2008 Jul;90(7):847-51. doi: 10.1302/0301-620X.90B7.20213. PMID 18591590
- [Background] Toms AP, Marshall TJ, Cahir J, Darrah C, Nolan J, Donell ST, Barker T, Tucker JK. MRI of early symptomatic metal-on-metal total hip arthroplasty: a retrospective review of radiological findings in 20 hips. Clin Radiol. 2008 Jan;63(1):49-58. doi: 10.1016/j.crad.2007.07.012. Epub 2007 Oct 24. PMID 18068790